CLINICAL TRIAL: NCT00353496
Title: Phase III, Randomised, Double-blind, Stratified Comparative, Placebo Controlled, Parallel Group, Multi-centre Study to Assess the Effect of Deep Subcutaneous Injections of Lanreotide Autogel 120mg Administered Every 28 Days on Tumour Progression Free Survival in Patients With Non-functioning Entero-pancreatic Endocrine Tumour
Brief Title: Study of Lanreotide Autogel in Non-functioning Entero-pancreatic Endocrine Tumours
Acronym: CLARINET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-55-52030-726; 2005-004904-35 (EudraCT Number)
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Endocrine Tumors
Keywords: Non functioning entero-pancreatic tumours
MeSH Terms: interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- lanreotide (Autogel formulation) (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — 120mg administered via deep subcutaneous injection every 28 days for a maximum period of 96 weeks.
  Arms: lanreotide (Autogel formulation)
Drug: Placebo — Saline solution 0.9% administered via deep subcutaneous injection every 28 days for a maximum period of 96 weeks.
  Arms: Placebo

SUMMARY:
The study will compare the difference between lanreotide Autogel and placebo on progression free survival in patients who have an endocrine tumour in the pancreas or intestines.

ELIGIBILITY:
Inclusion Criteria:

* Endocrine tumour in the intestine or pancreas and with locally advanced or metastatic disease
* No hormone related symptoms
* Well or moderately differentiated tumour confirmed by histology
* Tumour lesions which are measurable by a CT or MRI scan

Exclusion Criteria:

* Previously treated with a somatostatin analogue unless more than 6 months ago and given for no more than 15 days
* Treated within the last 6 months with interferon, chemoembolisation or chemotherapy or at any time with a radionuclide
* Had a previous cancer except basal cell carcinoma and/or in situ carcinoma of the cervix/uterus and/or patients treated with curative intent and free from disease for 5 years
* Pregnant or lactating
* Females must use adequate contraception during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2006-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Endocrinology, Study Director — Ipsen
Locations (71):
- United States (8):
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - University of Iowa, Iowa City, Iowa
  - The John Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- University Hospital, Vienna, Austria
- Belgium (3):
  - UZ Antwerpen, Antwerp
  - UCL Saint Luc, Brussels
  - UZ Gent, Ghent
- Czechia (3):
  - Fakultni nemocnice Na, Bulovce, Prague
  - Fekultni nemocnice Olomouc, Olomouc
  - General faculty, Prague
- Denmark (2):
  - Sygehus Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (9):
  - Hôpital A. Paré, Boulogne-Billancourt
  - Hôpital Beaujon, Clichy
  - CAC Oscar Lambret, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHU la Timone, Marseille
  - Hôpital R. Debré, Reims
  - CHI Frejus St Raphael, Saint-Raphaël
  - Hôpital Rangueil, Toulouse
  - Unité de gastro enterologie IGR, Villejuif
- Germany (6):
  - Charite Hospital, Berlin
  - University Hospital, Erlangen
  - University Hospital, Lübeck
  - Gutenberg University Hospital, Mainz
  - University Hospital, München
  - Lukas Hospital, Neuss
- India (2):
  - Global Hospital, Hyderabad
  - Tata Memorial Hospital, Mumbai
- Italy (6):
  - Centro di Refierimiento Oncologica, Aviano
  - Azienda Malpighi, Bologna
  - INSCT, Milan
  - University of Naples, Naples
  - Hospital S. Chiara, Pisa
  - Azienda San Giovanni Battista, Torino
- Netherlands (3):
  - UMC Gronigen, Gronigen
  - Erasmu MC, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (6):
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej - Curie, oddzial w Gliwicach, Zaklad Medycyny Nuklearnej i Endokrynologii Onkologicznej ul., Gliwice
  - Katedra i Klinika Endokrynologii Przemiany Materii i Chorob Wewnetrznych Uniwersytetu Medycznego w Poznaniu, Poznan
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Katedra i Klinika Chorob Wewnetrznych I Endokrynologii ul. Banacha 1 a, Warsaw
  - Szpital Bielanski im. Ks. Jerzego Popieluszki, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Klinika Endokrynologii Centrum Medycznego Ksztalcenia Podyplomowego, Warsaw
  - Zaklad Diagnosttyki Radiologicznej, Centralny Szpital Klincny, Ministrerstwa Spraw Wewnetrznych i Administratracji w Warzawie, Warsaw
  - Silesian Medical University, Zabrze
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava, Slovakia
  - Vychodoslovensky onkologicky ustav, Rastislavova, Slovakia
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Institut Catala Oncologia, Barcelona
  - Hospital G. Maranon, Madrid
  - Hospital La Paz, Madrid
  - Hospital Nuestra Senora de la Candelaria, Santa Cruz de Tenerife
- Sweden (3):
  - Sahlgrenska Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
  - University Hospital, Uppsala
- United Kingdom (12):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal Victoria Hospital, Belfast
  - University Hospital Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Free Hospital, London
  - St Bartholomew's Hospital, London
  - QMC, Nottingham
  - Churchill Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Derived] Caplin ME, Pavel M, Phan AT, Cwikla JB, Sedlackova E, Thanh XT, Wolin EM, Ruszniewski P; CLARINET Investigators. Lanreotide autogel/depot in advanced enteropancreatic neuroendocrine tumours: final results of the CLARINET open-label extension study. Endocrine. 2021 Feb;71(2):502-513. doi: 10.1007/s12020-020-02475-2. Epub 2020 Oct 14. PMID 33052555
- [Derived] Lybaert W, Van Hul E, Woestenborghs H. Long-term disease control of a pancreatic neuroendocrine tumor with lanreotide autogel((R)): a case report. Case Rep Oncol. 2014 Sep 26;7(3):673-80. doi: 10.1159/000368207. eCollection 2014 Sep. PMID 25408662
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2023/05/05101856/CLARINET-Clinical-Lay-summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 264 subjects were screened at 48 investigational sites in 14 countries (Austria, Belgium, Czech Republic, Denmark, France, Germany, India, Italy, Poland, Slovakia, Spain, Sweden, United Kingdom and the United States of America). 204 subjects were randomised to receive study treatment in the Intent to treat (ITT) population.
Period: Overall Study
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Started | 101 | 103
Completed | 85 (Patients who completed specified assessments or met primary efficacy endpoint criteria for an event.) | 86
Not Completed | 16 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 6 | 9
Not completed — Not otherwise specified | 4 | 2

BASELINE CHARACTERISTICS:
Population: Analysis based on intent-to-treat (ITT) population comprised of 204 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanreotide (Autogel Formulation) | Placebo | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 62 (11) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 53 | 54 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 97 | 96 | 193
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Time since diagnosis [Mean (Standard Deviation); unit: months] — Time relative to baseline visit (Week 1).
  months | 32.6 (46.1) | 34.4 (41.4) | 33.5 (43.7)
Neuroendocrine tumour (NET) origin [Number; unit: participants] — Primary tumour characteristics.
  participants
    Pancreas | 42 | 49 | 91
    Midgut | 33 | 40 | 73
    Hindgut | 11 | 3 | 14
    Unknown/Other | 15 | 11 | 26
Chromogranin A [Number; unit: participants] — Chromogranin A is an NET marker. ULN: upper limit of normal.
  participants
    ≤1 × ULN | 33 | 34 | 67
    1-2 × ULN | 25 | 18 | 43
    >2 × ULN | 41 | 48 | 89
    Unknown | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time from randomization to first documentation of disease progression, or death. Disease progression centrally assessed using Response Evaluation Criteria in Solid Tumours (RECIST) v1.0
Time Frame: From randomisation up to the last tumour assessment (scheduled at 96 weeks). Radiological scans were performed every 12 weeks during the first year and every 24 weeks during the second year
Population: Analysis based on the intent-to-treat (ITT) population which comprised 204 randomised subjects.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Lanreotide (Autogel Formulation): lanreotide (Autogel formulation): 120mg administered via deep subcutaneous injection every 28 days for a maximum period of 2 years.
- Placebo: Placebo: Saline solution 0.9% administered via deep subcutaneous injection every 28 days for a maximum period of 2 years.
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Number analyzed (Participants) | 101 | 103
Weeks | NA [NA to NA] — Not available as median not reached during the 96 week fixed duration study. | 72 [48.6 to 96.0]
Statistical Analysis 1: Comparison: Lanreotide (Autogel Formulation) vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank — No p-value adjustment for multiple comparisons; The log rank test was stratified according to progression status at baseline and prior therapy; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.30 to 0.73]

2. Secondary Outcome: Percentage of Patients Alive & Without Disease Progression
Description: Percentage of patients still ongoing (or completing at Week 96) without centrally assessed disease progression or death at Weeks 48 and 96.
Time Frame: Week 48 & 96
Population: Analysis based on the intent-to-treat (ITT) population which comprised 204 randomised subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Number analyzed (Participants) | 101 | 103
Percentage of participants
  Week 48 | 66 | 49
  Week 96 | 53 | 25

3. Secondary Outcome: Pharmacokinetic Profile of Lanreotide
Description: Pharmacokinetic Profile of Lanreotide assessed by mean serum concentration at specified timepoints
Time Frame: Week 4, 12, 24, 36, 48, 72, 96
Population: Analysis based on the intent-to-treat (ITT) population which comprised 101 randomised subjects who received lanreotide
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanreotide (Autogel Formulation)
Number analyzed (Participants) | 101
ng/mL
  At Week 4 predose (n=81) | 2.5 (0.46)
  At Week 12 predose (n=87) | 5.0 (0.42)
  At Week 24 predose (n=74) | 6.1 (0.44)
  At Week 36 predose (n=67) | 6.2 (0.39)
  At Week 48 predose (n=62) | 6.6 (0.45)
  At Week 72 predose (n=52) | 6.8 (0.44)
  At Week 96 predose (n=48) | 6.6 (0.39)

4. Secondary Outcome: Change in the Global Health Status Quality of Life Assessment
Description: Transformed scores from European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire responses (QLQ)-C30. Questionnaire response scores range from 0 to 100. Higher scores indicate best possible Quality of Life.
Time Frame: Week 12 to Week 96 (last visit)
Population: Analysis based on the intent-to-treat (ITT) population which comprised 193 randomised subjects with valid assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Number analyzed (Participants) | 95 | 98
score on a scale | -5.2 (3.7) | -4.9 (3.7)

5. Secondary Outcome: Percentage of Patients With a Greater Than or Equal to 50% Decrease in Plasma Chromogranin A (CgA) Levels
Time Frame: Week 12 to Week 96 (last visit)
Population: Analysis based on the subgroup of subjects with an elevated plasma CgA values. Subjects with a gastrinoma were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Number analyzed (Participants) | 64 | 64
percentage of participants | 42.2 | 4.7

6. Secondary Outcome: Percentage of Patients Still Alive Based on Available Overall Survival Data
Description: Overall survival defined as the time from randomisation to death due to any cause. Subjects were followed for overall survival beyond study completion/withdrawal via annual telephone contact until the last subject completed the study.
Time Frame: Randomisation to death or last visit, up to 321 weeks
Population: Analysis based on the intent-to-treat (ITT) population which comprised 204 randomised subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Number analyzed (Participants) | 101 | 103
percentage of participants | 84 | 77

ADVERSE EVENTS:
Time Frame: Total exposure to treatment was 138.0 subject years for lanreotide vs 123.6 subject years for placebo.
Arm/Group | Lanreotide (Autogel Formulation) | Placebo
Serious Adverse Events (participants affected / at risk) | 25/101 | 32/103
Other Adverse Events (participants affected / at risk) | 88/101 | 92/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide (Autogel Formulation) (N=101) | Placebo (N=103)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide (Autogel Formulation) (N=101) | Placebo (N=103)
Abdominal discomfort (Gastrointestinal disorders) | 5 (8) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 23 (32) | 18 (34)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 9 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (15) | 10 (11)
Asthenia (General disorders) | 8 (8) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 11 (11)
Cholelithiasis (Hepatobiliary disorders) | 15 (16) | 7 (7)
Constipation (Gastrointestinal disorders) | 11 (13) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (8)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 9 (9) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 35 (57) | 37 (75)
Dizziness (Nervous system disorders) | 9 (12) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (2)
Fatigue (General disorders) | 11 (15) | 16 (18)
Flatulence (Gastrointestinal disorders) | 12 (13) | 9 (12)
Flushing (Vascular disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 16 (19) | 11 (19)
Hypertension (Vascular disorders) | 13 (16) | 5 (5)
Injection site pain (General disorders) | 8 (30) | 4 (10)
Lethargy (Nervous system disorders) | 5 (13) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (6)
Nasopharyngitis (Infections and infestations) | 9 (10) | 17 (23)
Nausea (Gastrointestinal disorders) | 15 (28) | 13 (22)
Oedema peripheral (General disorders) | 5 (5) | 7 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Pancreatic enzymes decreased (Investigations) | 6 (7) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (17)
Pyrexia (General disorders) | 4 (6) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 8 (13) | 11 (13)
Vomiting (Gastrointestinal disorders) | 17 (21) | 10 (28)
Weight decreased (Investigations) | 9 (9) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No